CLINICAL TRIAL: NCT03974464
Title: Value of Copeptin and the S-100b Protein Assay in Ruling Out the Diagnosis of Stroke-induced Dizziness Pattern in Emergency Departments
Brief Title: Copeptin and the S-100b Protein in Stroke
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: vertigo
Record Dates: First submitted 2019-05-07; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Vertigo, Peripheral; Vertigo, Brain Stem; Vertigo; Central; Vertigo; Cerebral
Keywords: vertigo; stroke; copeptin; S-100b protein; biomarkers
MeSH Terms: conditions — Vertigo; Stroke; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PS100 concentrations were measured on serum samples by electro-chemiluminescence assay (Roche, Mannheim, Germany). Copeptin concentrations were measured on serum samples by the Kryptor method (Thermo Scientific, Hennigsdorf, Germany)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: copeptin, PS100 — Age, sex and time between dizziness onset and ED visit were collected using Resurgences® software. PS100 concentrations were measured on serum samples by electro-chemiluminescence assay. Copeptin concentrations were measured on serum samples by the Kryptor method. The positivity threshold for copeptin was set at strictly above 10 pmol/L and that of PS100 was set at strictly above 0.105 μmol/L.
  And after, we compared results with results of brain imaging: Magnetic Resonance Imaging alone, CT scan alone or both. Depending on clinical presentation, the imaging tests were performed during ED stay, during hospitalization or externally. Presence or absence of stroke was established on diffusion-weighted brain MRI . In case of normal contrast CT alone, a specialized opinion should exclude the need for diffusion-weighted MRI according to clinical presentation.

SUMMARY:
This study evaluated the value of using copetin and protein S 100 b to eliminate the diagnosis of stroke in patients presenting with vertigo in emergency departments. All patients benefited from the S 100b protein assay, copeptin and brain MRI.

DETAILED DESCRIPTION:
Vertigo is a frequent reason for visiting emergency departments. Differentiating stroke from other causes is challenging for physicians. The role of biomarkers has been poorly assessed. Evaluators evaluated whether copeptin and S100b protein assessment, alone or in combination, could rule out stroke in patients visiting emergency departments for vertigo.

Evaluators included patients visiting the adult emergency departments of a French university hospital for a new episode of vertigo evolving for less than 72 hours. All patients underwent standardized physical examination (HINT [Head Impulse test, Nystagmus, test of skew deviation] maneuvers), copeptin and S-100b protein measurement and injected brain imaging. Stroke diagnosis involved diffusion-weighted magnetic resonance imaging or, if not available, neurological examination and contrast brain CT scan compatible with the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* We included patients 18 years of age or older, visiting the ED for a new episode of dizziness evolving less than 72 hours and having given written consent to participate in the study

Exclusion Criteria:

* Patients without brain imaging (diffusion-weighted magnetic resonance imaging (MRI) or contrast CT scan compatible with the diagnosis) were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred and fifty-one patients were included, of whom 16 were secondarily excluded (lost to follow-up n=1, missing biomarkers n=9, missing MRI n=6)(Figure 1). A majority of the remaining 135 patients were women (n=79, 59%) with an average age of 62 years . Specialized advice on the origin of dizziness was sought from ENT and/or neurologist in 102 (76%) of cases. Patients received brain diffusion-weighted MRI alone in 74 cases, contrast brain CT alone in 11 cases and a combination of MRI and CT in 50 cases. In 122 patients (90%), vertigo was not related to stroke.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Show that the negativity of S-100b protein and copeptin eliminates stroke in the face of vertigo | 1 hour
  negative predictive value of the S-100b protein and copeptin combination

IPD SHARING:
Plan to Share IPD: No